CLINICAL TRIAL: NCT01093404
Title: Thrombus Aspiration in ST- Elevation Myocardial Infarction in Scandinavia
Brief Title: Thrombus Aspiration in Myocardial Infarction
Acronym: TASTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Ole Frobert, MD, PhD, MD, PhD, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCAAR-001
Record Dates: First submitted 2010-03-22; First posted 2010-03-25 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myocardial Infarction
Keywords: Heart disease; Myocardial infarction; Angioplasty; Thrombus aspiration
MeSH Terms: conditions — Heart Diseases; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thrombus aspiration (Experimental): Thrombus aspiration is then followed by standard balloon angioplasty (PCI).
  Interventions: Procedure: Thrombus aspiration
- Standard balloon angioplasty (PCI) (Active Comparator)
  Interventions: Procedure: Thrombus aspiration

INTERVENTIONS:
Procedure: Thrombus aspiration — Aspiration of thrombus material before angioplasty

SUMMARY:
Treatment of myocardial infarction (blood clot in the arteries of the heart) has improved after introduction of 24/7 balloon angioplasty to open the blocked artery. However, the clot itself is not routinely removed but recent data in smaller trials indicate that this might improve recovery and prognosis. In this multicenter study of 5000 patients referred to Scandinavian hospitals for myocardial infarction the investigators test the hypothesis that patients randomized to treatment with thrombus aspiration (removing the blood clot by manual suction) before conventional angioplasty will have a reduced risk of death, fewer rehospitalisations, fewer new myocardial infarctions, reduced risk of heart failure, better coronary artery flow after angioplasty and greater reduction of infarct size compared to patients randomized to conventional angioplasty alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ST-segment elevation myocardial infarction
* Correspondence between ECG findings and culprit artery pathoanatomy
* A minimum of 50% stenosis in culprit artery by visual estimate
* Possibility to perform thrombus aspiration

Exclusion Criteria:

* Need for emergency coronary artery bypass grafting
* Inability to provide informed consent
* Age below 18 years
* Previous randomization in the TASTE trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7243 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
All-cause death | 30 days
  Death from any cause will be registered via national registries during the first 30 days after study inclusion.

SECONDARY OUTCOMES:
Time to re-hospitalization with nonfatal reinfarction, heart failure and target vessel revascularization | 30 days to 10 years
Time to all-cause death or new myocardial infarction (first occurring) or in hospital treatment for heart failure | 30 days to 10 years
Time to acute coronary occlusion, stent thrombosis and restenosis in treated lesions | 1 year
Length of hospital stay | 1 month
TIMI-flow grade | 3 hours
  TIMI-flow, or Thrombolysis in Myocardial Infarction grading of flow is a semiquantitative method to assess coronary artery flow following balloon angioplasty.
All-cause death | 1 year to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ole Fröbert, MD, PhD, Principal Investigator — Region Örebro County
Locations (29):
- Skejby Hospital, Aarhus University Hospital, Aarhus, Denmark
- Landspitali University Hospital, Reykjavik, Iceland
- Sweden (27):
  - Södra Älvsborgs sjukhus, Borås
  - Mälarsjukhuset, Eskilstuna
  - Falu lasarett, Falun
  - Gävle sjukhus, Gävle
  - Sahlgrenska sjukhuset, Gothenburg
  - Östra sjukhuset, Gothenburg
  - Hallands sjukhus, Halmstad
  - Helsingborgs lasarett, Helsingborg
  - Länssjukhuset Ryhov, Jönköping
  - Länssjukhuset, Kalmar
  - Blekingesjukhuset, Karlskrona
  - Svensk PCI AB, Centralsjukhuset, Karlstad
  - Centralsjukhuset, Kristianstad
  - Universitetssjukhuset, Linköping
  - Sunderby sjukhus, Luleå
  - Lund University Hospital, Lund
  - Skånes universitetssjukhus, Malmo
  - Örebro University Hospital, Örebro
  - Karolinska universitetssjukhuset, Solna
  - Danderyds sjukhus, Stockholm
  - S:t Görans sjukhus, Stockholm
  - Södersjukhuset, Stockholm
  - Länssjukhuset, Sundsvall
  - Norra Älvsborgs länssjukhus, Trollhättan
  - Universitetssjukhuset, Umeå
  - Uppsala University Hospital, Uppsala
  - Centrallasarettet, Västerås

REFERENCES:
- [Derived] Calais F, Lagerqvist B, Leppert J, James SK, Frobert O. Thrombus aspiration in patients with large anterior myocardial infarction: A Thrombus Aspiration in ST-Elevation myocardial infarction in Scandinavia trial substudy. Am Heart J. 2016 Feb;172:129-34. doi: 10.1016/j.ahj.2015.11.012. Epub 2015 Nov 22. PMID 26856224
- [Derived] Frobert O, Calais F, James SK, Lagerqvist B. ST-elevation myocardial infarction, thrombus aspiration, and different invasive strategies. A TASTE trial substudy. J Am Heart Assoc. 2015 Jun 15;4(6):e001755. doi: 10.1161/JAHA.114.001755. PMID 26077585
- [Derived] Lagerqvist B, Frobert O, Olivecrona GK, Gudnason T, Maeng M, Alstrom P, Andersson J, Calais F, Carlsson J, Collste O, Gotberg M, Hardhammar P, Ioanes D, Kallryd A, Linder R, Lundin A, Odenstedt J, Omerovic E, Puskar V, Todt T, Zelleroth E, Ostlund O, James SK. Outcomes 1 year after thrombus aspiration for myocardial infarction. N Engl J Med. 2014 Sep 18;371(12):1111-20. doi: 10.1056/NEJMoa1405707. Epub 2014 Sep 1. PMID 25176395
- [Derived] Frobert O, Lagerqvist B, Olivecrona GK, Omerovic E, Gudnason T, Maeng M, Aasa M, Angeras O, Calais F, Danielewicz M, Erlinge D, Hellsten L, Jensen U, Johansson AC, Karegren A, Nilsson J, Robertson L, Sandhall L, Sjogren I, Ostlund O, Harnek J, James SK; TASTE Trial. Thrombus aspiration during ST-segment elevation myocardial infarction. N Engl J Med. 2013 Oct 24;369(17):1587-97. doi: 10.1056/NEJMoa1308789. Epub 2013 Aug 31. PMID 23991656
- [Derived] Frobert O, Lagerqvist B, Gudnason T, Thuesen L, Svensson R, Olivecrona GK, James SK. Thrombus Aspiration in ST-Elevation myocardial infarction in Scandinavia (TASTE trial). A multicenter, prospective, randomized, controlled clinical registry trial based on the Swedish angiography and angioplasty registry (SCAAR) platform. Study design and rationale. Am Heart J. 2010 Dec;160(6):1042-8. doi: 10.1016/j.ahj.2010.08.040. PMID 21146656
- [Derived] Frobert O, Lagerqvist B, Kreutzer M, Olivecrona GK, James SK. Thrombus aspiration in ST-elevation myocardial infarction in Sweden: a short report on real world outcome. Int J Cardiol. 2010 Dec 3;145(3):572-3. doi: 10.1016/j.ijcard.2010.05.044. Epub 2010 Jun 13. No abstract available. PMID 20550973
- See also: Related Info — http://www.ucr.uu.se/scaar/